CLINICAL TRIAL: NCT05144256
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Mitapivat in Pediatric Subjects With Pyruvate Kinase Deficiency Who Are Regularly Transfused, Followed by a 5-Year Open-label Extension Period
Brief Title: A Study to Evaluate the Efficacy and Safety of Mitapivat in Pediatric Participants With Pyruvate Kinase Deficiency (PKD) Who Are Regularly Transfused, Followed by a 5-Year Extension Period
Acronym: ACTIVATE-KidsT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG348-C-022; 2021-003265-36 (EudraCT Number); 2024-515024-37-00 (EU CTIS Number)
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Pyruvate Kinase Deficiency; Pediatric Hemolytic Anemia
Keywords: Anemia; Hematologic Diseases; Metabolic Diseases; Mitapivat; AG-348; ACTIVATE-KidsT; PK Deficiency
MeSH Terms: conditions — Anemia; Hematologic Diseases; Metabolic Diseases; Pyruvate Kinase Deficiency of Red Cells | interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mitapivat (Experimental): For participants randomized to receive mitapivat, dosing occurs orally twice daily (BID), and is based on age and weight. Dosing is optimized through 2 potential sequential increases in dose levels (1-5 mg, 4-20 mg and 10-50 mg) at Week 4 and Week 8, and aims to achieve the adult-equivalent exposure at 5, 20, and 50 mg. Following titration, participants remain on their individually optimized dose during the remainder of the Double-blind (DB) Period for 24 weeks. After the DB period, participants will enter an Open-label Extension (OLE) Period. To preserve blinding of treatment allocation, participants will continue mitapivat at their optimized dose and undergo mock titration with placebo for 8 weeks. At the conclusion of 8 weeks, participants may continue receiving mitapivat in the OLE Period for up to 262 weeks (including up to 2 weeks of dose taper).
  Interventions: Drug: Mitapivat; Drug: Mitapivat-matching placebo
- Placebo (Placebo Comparator): For participants randomized to receive matched placebo, dosing is identical to that described above for mitapivat. Following the initial dose titration period, participants remain on their individually optimized dose during the remainder of the DB period for 32 weeks. After the DB period, participants will enter an OLE period. To preserve blinding of treatment allocation, participants will continue placebo at their optimized dose and undergo mitapivat dose optimization through 2 potential sequential increases in dose levels (1-5 mg, 4-20 mg and 10-50 mg) at Week 4 and Week 8 of the OLE Period, and aims to achieve the adult-equivalent exposure at 5, 20, and 50 mg. At the conclusion of 8 weeks, participants may continue receiving mitapivat in the OLE Period for up to 262 weeks (including up to 2 weeks of dose taper).
  Interventions: Drug: Mitapivat; Drug: Mitapivat-matching placebo

INTERVENTIONS:
Drug: Mitapivat — Tablets or granules
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate
Drug: Mitapivat-matching placebo — Tablets or granules

SUMMARY:
ACTIVATE-KidsT (AG348-C-022) is a multicenter study designed to evaluate the efficacy and safety of treatment with mitapivat compared with placebo in pediatric participants with pyruvate kinase deficiency (PK deficiency) who are regularly receiving blood transfusions. Participants will be randomized 2:1 to receive either mitapivat or matching placebo. Randomization will be stratified by age (1 to < 6 years, 6 to < 12 years, 12 to < 18 years) and splenectomy status. Participants will be dosed by age and weight during a double-blind period consisting of an 8-week dose titration period followed by a 24-week fixed-dose period. Participants who complete the double-blind period will be eligible to receive mitapivat in the open-label extension (OLE) period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the participant, or the participant's legally authorized representative, parent(s), or legal guardian, and the participant's assent, where applicable (informed consent/assent) must be obtained before any study-related procedures are conducted, and participants must be willing to comply with all study procedures for the duration of the study;
* Aged 1 to <18 years. Participants between 12 and 24 months of age must weigh a minimum of 7 kilograms (kg);
* Clinical laboratory confirmation of pyruvate kinase deficiency (PKD), defined as documented presence of at least 2 mutant alleles in the pyruvate kinase L/R (PKLR) gene, of which at least 1 is a missense mutation, as determined per the genotyping performed by the study central genotyping laboratory;
* Six to 26 transfusion episodes in the 52-week period before providing informed consent/assent;
* Have complete records of transfusion history for the 52 weeks before providing informed consent/assent, defined as having all the following available: (1) all the transfusion dates, (2) the RBC transfusion volume (milliliters and/or number of units) for all the transfusions, and (3) hemoglobin concentrations within 1 week before transfusion for at least 80% of the transfusions;
* Receiving folic acid supplementation as part of routine clinical care for at least 21 days before administration of the first dose of study drug, to be continued during study participation;
* Female participants who have attained menarche and/or breast development in Tanner Stage 2 must be abstinent of sexual activities that may induce pregnancy as part of their usual lifestyle, or agree to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of informed consent/assent, throughout the study, and for 28 days after the last dose of study drug (including the time required to dose taper). The second form of contraception can include an acceptable barrier method.

Exclusion Criteria:

* Pregnant or breastfeeding;
* Homozygous for the R479H mutation or have 2 nonmissense mutations, without the presence of another missense mutation, in the PKLR gene as determined per the genotyping performed by the study central genotyping laboratory;
* History of malignancy;
* History of active and/or uncontrolled cardiac or pulmonary disease or clinically relevant QT prolongation within 6 months before providing informed consent/assent;
* Hepatobiliary disorders including, but not limited to:

  * Liver disease with histopathological evidence of cirrhosis or severe fibrosis;
  * Clinically symptomatic cholelithiasis or cholecystitis (participants with prior cholecystectomy are eligible);
  * History of drug-induced cholestatic hepatitis;
  * Aspartate aminotransferase >2.5×upper limit of normal (ULN) (unless due to hemolysis and/or hepatic iron deposition) and alanine aminotransferase >2.5×ULN (unless due to hepatic iron deposition);
* Renal dysfunction as defined by an estimated glomerular filtration rate <60 milliliters per minute (mL/min)/1.73 m^2;
* Nonfasting triglycerides >440 milligrams per deciliter (mg/dL) (5 millimoles per liter [mmol/L]);
* Active uncontrolled infection requiring systemic antimicrobial therapy;
* Participants with known active hepatitis B or hepatitis C virus infection;
* Participants with known human immunodeficiency virus (HIV) infection;
* History of major surgery (including splenectomy) ≤6 months before providing informed consent/assent and/or planning on undergoing a major surgical procedure during the screening or double-blind period;
* Current enrollment or past participation (within 90 days before the first dose of study drug or a time frame equivalent to 5 half-lives of the investigational study drug, whichever is longer) in any other clinical study involving an investigational study drug or device;
* Prior exposure to gene therapy, or bone marrow or stem cell transplantation;
* Currently receiving hematopoietic stimulating agents; the last dose must have been administered at least 28 days or a time frame equivalent to 5 half-lives (whichever is longer) before randomization;
* Receiving products that are strong inhibitors of CYP3A4/5 that have not been stopped for ≥5 days or a time frame equivalent to 5 half-lives (whichever is longer), or strong inducers of CYP3A4 that have not been stopped for ≥28 days or a time frame equivalent to 5 half-lives (whichever is longer), before randomization;
* Receiving anabolic steroids, including testosterone preparations, that have not been stopped for at least 28 days before randomization;
* Known allergy, or other contraindication, to mitapivat or its excipients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, Opadry® II Blue [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and Food, Drug, and Cosmetics blue dye number 2 (FD&C Blue #2)], Opadry® II White [hypromellose, titanium dioxide, lactose monohydrate, and triacetin], and magnesium stearate);
* Any medical, hematologic, psychological, or behavioral condition(s) or prior or current therapy that, in the opinion of the Investigator, may confer an unacceptable risk to participating in the study and/or could confound the interpretation of the study data; also included are:

  * Participants who are institutionalized by regulatory or court order.
  * Participants with any condition(s) that could create undue influence (including but not limited to incarceration, involuntary psychiatric confinement, and financial or familial affiliation with the Investigator or Sponsor).
* Receiving a pyruvate kinase activator that has not been stopped for ≥52 weeks before providing informed consent/assent.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Transfusion Reduction Response (TRR) | Week 9 to Week 32
  TRR is defined as ≥33% reduction in total red blood cell (RBC) transfusion volume from Week 9 through Week 32 of the double-blind period, normalized by weight and actual study drug duration compared with the historical transfusion volume, standardized by weight, and to 24 weeks.

SECONDARY OUTCOMES:
Percentage of Participants With Transfusion-free Response | Week 9 to Week 32
  Transfusion-free response is defined as achievement of 0 transfusions administered from Week 9 through Week 32 of the double-blind period.
Change in the Number of Transfusion Episodes | Week 9 to Week 32
  The change in the number of transfusion episodes from Week 9 through Week 32 of the double-blind period compared with the historical number of transfusion episodes standardized to 24 weeks.
Percentage Change in Weight-normalized and Study Treatment Duration-normalized Total Transfusion Volume | Week 9 to Week 32
  The percentage change in weight-normalized and study treatment duration-normalized total transfusion volume from Week 9 through Week 32 of the double-blind period will be compared with the historical transfusion volume standardized by weight and to 24 weeks.
Percentage of Participants With Normal Hemoglobin (Hb) Response | Week 9 to Week 32
  Normal Hb response is defined as achievement of Hb concentrations in the normal range at least once, 8 weeks or more after a transfusion during Week 9 through Week 32 of the double-blind period.
Change From Baseline in Estradiol Concentration | Baseline up to Week 298
Change From Baseline in Estrone Concentration | Baseline up to Week 298
Change From Baseline in Total Testosterone Concentration | Baseline up to Week 298
Change From Baseline in Free Testosterone Concentration in Participants ≥7 Years of Age or Tanner Stage ≥2 (Whichever Occurs First) | Baseline up to Week 298
Change From Baseline in Luteinizing Hormone Concentration in Participants ≥6 Years of Age | Baseline up to Week 298
Change From Baseline in Sexual Maturity Rating with Tanner Stage | Baseline up to Week 298
  Tanner Stage 1 corresponds to the prepubertal form, with progression to Tanner Stage 5, the final adult form.
Percentage Number of Female Participants With Development of Ovarian Cysts | Baseline up to Week 298
Change From Baseline in the Size of Ovarian Cysts in Female Participants | Baseline up to Week 298
Change From Baseline in Height-for-age Z-score | Baseline up to Week 298
Change From Baseline in Weight-for-age Z-score | Baseline up to Week 298
Change From Baseline in Body Mass Index (BMI)-for-age Z-score | Baseline up to Week 298
Change From Baseline in Bone Mineral Density (BMD) Z-score | Baseline up to Week 298
Change from Baseline in Serum Iron Concentration | Baseline up to Week 292
Change from Baseline in Serum Ferritin Concentration | Baseline up to Week 292
Change from Baseline in Total Iron-binding Capacity | Baseline up to Week 292
Change from Baseline in Transferrin/Transferrin Saturation | Baseline up to Week 292
Change from Baseline in Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale | Baseline up to Week 292
  The PedsQL multidimensional fatigue scale yields a total score from age-appropriate validated questionnaire that asks for perceived fatigue within the domains of 'General', 'Sleep/Rest' and 'Cognitive'. Each domain consists of 6 questions that are rated from 0 to 4 (therefore total score can range from 0 to 72). A higher total score indicates greater fatigue (i.e., worse outcome).
Change from Baseline in PedsQL Generic Core Scale (GCS) | Baseline up to Week 292
  PedsQL GCS is designed to measure health-related quality of life in pediatric participants and adolescents (2 to 18 years of age). It encompasses 4 dimensions of functioning (physical [8 items], emotional [5 items], social [5 items], school [3 items]). Age groups: Toddler (2-4 years), Young pediatric (5-7 years), Pediatric (8-12 years), and Teens (13-17 years). Depending on the participant's age, the questionnaire may be completed by parent/caregiver as appropriate. For the Toddler group, the PedsQL GCS consist of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consist of 23 items, with a 3-point Likert scale (0, 2, 4) for the young pediatric, and a 5-point Likert scale for the pediatric and teens groups. Scores are transformed on a scale from 0 to 100 where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Population Pharmacokinetic (PK) Model Parameter Estimate: Maximum Plasma Concentration (Cmax) of Mitapivat | Weeks 2, 8, 12, and 16
Population PK Model Parameter Estimate: Area Under the Concentration-time Curve (AUC) Derived From Plasma Concentrations of Mitapivat | Weeks 2, 8, 12, and 16
Concentration at Steady State (Css) of Mitapivat | Week 16: 6 and 8 hours postdose
Trough Concentration (Ctrough) of Mitapivat | Week 8: ≤30 minutes predose; Week 12: ≤30 minutes predose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (22):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford Medicine, Palo Alto, California
  - Children's Healthcare of Atlanta - Emory, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Cure 4 the Kids Foundation, A Division of Roseman University of Health Sciences, Las Vegas, Nevada
  - Weill Cornell Medical College, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Comprehensive Hemophilia Care Clinic at CHEO (Children's Hospital Eastern Ontario), Ottawa, Ontario, Canada
- Fakultní Nemocnice Olomouc, Olomouc, Czechia
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Rigshospitalet, Copenhagen
- Charite - UB - CVK - Medizinische Klinik, Berlin, Germany
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinico Universitario Virgen de la Arrixaca, Madrid
- CHUV University Hospital of Lausanne, Lausanne, Canton of Bern, Switzerland
- Turkey (Türkiye) (3):
  - Ege University Faculty of Medicine, Izmir, Adana
  - Hacettepe University, Ankara
  - İstanbul Üniversitesi Tıp Fakültesi [Istanbul University Faculty of Medicine] Çocuk Sağlığı Enstitüsü [Institute of Child Health], Istanbul
- King's College Hospital NHS, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No